CLINICAL TRIAL: NCT04239469
Title: Phase II Clinical Trial, Use of KL16-012 in Women With Fibromyalgia Refractary to Conventional Treatment.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Knop Laboratorios (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PC003DT
Record Dates: First submitted 2020-01-05; First posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Fibromyalgia; Cannabis
Keywords: cannabis; fibromyalgia; phytocannabinoids; cannabinoid
MeSH Terms: conditions — Fibromyalgia; Marijuana Abuse

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KL16-012 (Active Comparator): Patients will use a liquid standardized extract of cannabis sativa. Each drop will contain 1 mg of THC and 0.45 mg of CBD. Administration will be sublingual, while dosing will begin at 3 drops per day and be escalated to 15 drops per day by week 5 according to an escalation chart.
  Interventions: Drug: KL16-012
- Placebo (Placebo Comparator): Patients will use a liquid placebo identical to the active principle in both appearance and taste.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: KL16-012 — Standardized cannabis sativa extract of THC and CBD, with each drop containing 1 mg of THC and 0.45 mg of CBD
  Other Names: Cannabiol
  Arms: KL16-012
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
A double blind randomized placebo controlled trial in 44 women with fibromyalgia and persistent symptoms in spite of use of conventional pharmacotherapy, will be performed in the city of Valparaiso. Patients will be randomized to either placebo or active principle and be followed for 3 months. Assesment of efficacy and safety will be done by measurement of changes in their Fibromyalgia Impact Questionnaire (FIQ) score, Insomnia Severity Index (ISI) score, pain Visual Analogue Scale (VAS) score, plasma cytokine levels and detection of adverse effects.

The active principle will be a standardized extract of cannabis sativa containing 1 milligram of tetrahydrocannabinol (THC) and 0.45 milligrams cannabidiol (CBD) per drop.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of fibromyalgia based on ACR 2010 criteria
* FIQ > 39 (refractary symptoms)
* Previous use of at least 2 conventional pharmacotherapies

Exclusion Criteria:

* History of substance use disorder
* History of major psychiatric or cardiovascular diseases
* Pregnancy
* Urine THC (+)

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2020-01-15 (Estimated); Primary Completion 2020-06-15 (Estimated); Study Completion 2020-09-15 (Estimated)

PRIMARY OUTCOMES:
Change in Fibromyalgia Impact Questionnaire (FIQ) score | Baseline to 12 weeks
  Numeric score validated in its spanish version, with scores ranging from 0 to 104 and higher values indicating worse symptoms.

SECONDARY OUTCOMES:
Change in Fibromyalgia Impact Questionnaire (FIQ) score | Baseline to 2 weeks
  Numeric score validated in its spanish version, with scores ranging from 0 to 104 and higher values indicating worse symptoms.
Change in Fibromyalgia Impact Questionnaire (FIQ) score | Baseline to 4 weeks
  Numeric score validated in its spanish version, with scores ranging from 0 to 104 and higher values indicating worse symptoms.
Change in Fibromyalgia Impact Questionnaire (FIQ) score | Baseline to 8 weeks
  Numeric score validated in its spanish version, with scores ranging from 0 to 104 and higher values indicating worse symptoms.
Change in Insomnia Severity Index (ISI) score | Baseline to 2 weeks
  Numeric score validated in its spanish version, with scores ranging from 0 to 28 and higher scores indicating worse insomnia.
Change in Insomnia Severity Index (ISI) score | Baseline to 4 weeks
  Numeric score validated in its spanish version, with scores ranging from 0 to 28 and higher scores indicating worse insomnia.
Change in Insomnia Severity Index (ISI) score | Baseline to 8 weeks
  Numeric score validated in its spanish version, with scores ranging from 0 to 28 and higher scores indicating worse insomnia.
Change in Insomnia Severity Index (ISI) score | Baseline to 12 weeks
  Numeric score validated in its spanish version, with scores ranging from 0 to 28 and higher scores indicating worse insomnia.
Change in pain Visual Analog Scale (VAS) score | Baseline to 2 weeks
  Numeric visual analog scale, with scores ranging from 0 to 10 and higher scores indicating worse pain.
Change in pain Visual Analog Scale (VAS) score | Baseline to 4 weeks
  Numeric visual analog scale, with scores ranging from 0 to 10 and higher scores indicating worse pain.
Change in pain Visual Analog Scale (VAS) score | Baseline to 8 weeks
  Numeric visual analog scale, with scores ranging from 0 to 10 and higher scores indicating worse pain.
Change in pain Visual Analog Scale (VAS) score | Baseline to 12 weeks
  Numeric visual analog scale, with scores ranging from 0 to 10 and higher scores indicating worse pain.
Changes in plasma cytokines | Baseline to 12 weeks
  Quantitative ELISA measurements of plasma levels of IL-6, IL-8, CXCL5, CXCL6, MCP-2, LAP TGFβ-1 and TNFα

IPD SHARING:
Plan to Share IPD: No